CLINICAL TRIAL: NCT00504140
Title: Phase II Study of Recombinant Interferon Alpha and Etoposide in Patients With Relapsed Osteosarcoma
Brief Title: Recombinant Interferon Alpha and Etoposide in Relapsed Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P96-221
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Interferon Alpha; IFN-; Roferon; Recombinant Interferon Alpha; Etoposide; VP-16
MeSH Terms: conditions — Osteosarcoma | interventions — Etoposide; Interferon-alpha; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interferon Alpha + Etoposide (Experimental): Interferon Alpha 5x10^6 mu/m^2 subcutaneously and Etoposide 100 mg/m^2 intravenously, both daily for 5 days
  Interventions: Drug: Etoposide; Drug: Interferon Alpha

INTERVENTIONS:
Drug: Etoposide — 100 mg/m^2 Intravenous Daily for 5 days, beginning one hour after IFN-alpha treatment.
  Other Names: VP-16
Drug: Interferon Alpha — 5x10^6 mu/m^2 Subcutaneously Daily for 5 Days
  Other Names: IFN-; Roferon

SUMMARY:
Primary Objectives:

1. To determine the efficacy of combining Interferon Alpha (IFN) with etoposide for the treatment of relapsed osteosarcoma.
2. To determine if IFN alters the plasma pharmacokinetics of etoposide.
3. To determine the toxicities of IFN and etoposide when administered together.
4. To determine IFN blood levels following combination therapy.

DETAILED DESCRIPTION:
Interferon Alpha (IFN)- will be given as a shot under the skin. One hour later, VP-16 will be infused through a catheter (tube) placed in a vein over 3 hours. The drugs will be given daily for 5 days. The treatment will be repeated every 3 - 4 weeks for up to 24 - 32 weeks (8 courses). The catheter will remain in place throughout treatment.

Patients who are candidates for surgery will first receive two courses of treatment. If the tumor gets worse or if severe side effects occur, treatment will be stopped, and the tumor will be removed right away. If the tumor responds well (begins to shrink or does not get worse) and severe side effects do not occur, the patient will receive six more courses of treatment after surgery.

Patients who are not candidates for surgery will receive two initial courses of treatment. If the tumor responds well and severe side effects do not occur, the patient will receive six more courses of treatment.

The treatment will be given in the outpatient department. Before treatment begins, the patient will have a health examination. Blood tests, a urine test, and heart tests will be given. X-rays, computed tomography (CT) scans, and a bone scan will be done. The location and size of all lesions will be recorded.

During treatment, patients will have a blood test every week. Before each course, a health examination, a urine test, and chest x-ray will be given and the size of all measurable cancer will be recorded. After the second course, the CT and bone scans will be repeated. All the tests will be repeated at the end of the study.

About 37 patients will be treated on the study at M. D. Anderson.

THIS IS AN INVESTIGATIONAL STUDY. IFN- and VP-16 are approved by the U.S. Food and Drug Administration for treating some types of cancer. Their use together against osteosarcoma is investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed relapsed osteosarcoma who have failed standard chemotherapy.
2. Age 5-70 years.
3. Life expectancy of at least 12 weeks and a Zubrod performance status of less than or equal to 2.
4. Patients must have measurable disease.
5. Adequate hematologic, coagulation, renal, and hepatic function.
6. No chemotherapy, immunotherapy, hormonal therapy or radiation therapy within 3 weeks of study entry.

Exclusion Criteria:

1. Patients who are likely to have significant systems because of rapidly progressive disease, ascites or hepatic metastasis.
2. Pregnant or lactating women.
3. Patients who have had more than one prior biologic response modifier.
4. Serious intercurrent illness, active infections, or central nervous system (CNS) disease.
5. Patients of childbearing potential, not practicing adequate contraception.
6. Significant cardiovascular disease.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1996-11; Primary Completion 2007-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Response when combining IFN with etoposide for the treatment of relapsed osteosarcoma. | Up to 24 - 32 weeks (8 courses of 3 - 4 weeks)
  Complete Response (CR): Disappearance of all evidence of tumor for at least one cycle; Lytic or mixed bone lesions improved by scan or shown some ossification by x-ray; and free of all symptoms of cancer. Partial Response (PR): 50% or > decrease in sum of product of diameters of all measured lesions persisting for at least one cycle or 4 weeks. No lesion may increase in size or new lesion appear. Minor Response (MR): Decrease in measurable lesion(s) too small or too brief to qualify as Partial Response.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenie S. Kleinerman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org